CLINICAL TRIAL: NCT01367353
Title: Characterization of Ovarian Cancer Stem Cell: Focus on Identification of Biomarker and Drug Resistance
Brief Title: Characterization of Ovarian Cancer Stem Cell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wen-Fang Cheng/Professor, National Taiwan Unviersity Hospital
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200902010R
Record Dates: First submitted 2010-12-10; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ovarian cancer (Experimental)
  Interventions: Procedure: surgery or debulking surgery

INTERVENTIONS:
Procedure: surgery or debulking surgery — surgery or debulking surgery

SUMMARY:
Specific aims: Identification and characterization of cancer stem cell-like population (cancer stem cells or cancer initiating cells) from primary tumor tissue, primary ascites and peripheral blood of ovarian cancer patients and genetically engineered mouse ovarian cancer cell lines.

Objectives: In the future, individualized therapy must incorporate analysis of the cancer stem cells or cancer initiating cells of ovarian cancer cells when designing therapeutic strategies for ovarian cancer patients.

Aims of this project:

1. Isolation and identification of cancer stem cell-like population (cancer stem cells or cancer initiating cells) from primary tumor tissue, primary ascites and peripheral blood of ovarian cancer patients
2. In vivo tumorigenicity assay will be performed to measure tumor formation from these cancer stem cell-like population when equal numbers were injected into the dorsal fat pad of nude mice.
3. To establish a standard protocol of stem cell-like population maintenance
4. Screening of potential specific biomarkers involved in these ovarian cancer stem cell-like population.

DETAILED DESCRIPTION:
Ovarian cancer has the highest mortality of all gynecological cancers, with an overall 5-year survival rate of only 30-40%. The incidence of ovarian cancer also increased in recent year in Taiwan, and it became a more and more important issue. The lack of symptoms, difficulties in early diagnosis, insufficient accurate tumor markers, and lack of information about ovarian tumor biology contribute to the poor prognosis in ovarian cancer patients. The prognostic factors for ovarian carcinomas include tumor stage, subtype of histology, grade of differentiation, the residual tumor after debulking surgery, and the response to chemotherapy. Especially the resistance to chemotherapy plays a great role in the prognosis of the patients. However, the current studies present an incomplete picture of the tumor biology of ovarian cancer. It will be quite helpful to clinical management if the investigators can examine the possible underlying mechanism of tumorigenesis and drug resistance.

Malignancy usually origins from the abnormal proliferate cells which accumulate several genetic or epigenetic aberrations. The most important key question is "What kind of cell could be the cancer cell?" Recent studies figure out there is "cancer-initiating cell" in the malignant tumor. Cancer-initiating cells organized self-renewing, anchorage-independent spheres and were reproducibly. Moreover, cancer-initiating cells were also capable of intraperitoneal tumorigenesis (demonstrating activity in their native microenvironment) and could serially propagate tumors in animals. Although the proportion of the cancer-initiating cells in the cancer tissue is very low, the characteristic abilities of cancer-initiating cells fulfill all currently accepted criteria for the existence of a subpopulation of tumor-initiating cells, and their specific detection and targeting could be highly valuable for therapy of tumor heterogeneity, uncontrolled proliferation, local invasion, distant metastasis and even resistance to current management including chemotherapy.

Some tumor initiating cells which have the properties of cancer stem cells have been isolated from leukemia, breast cancer, and brain tumor. Some potential cell markers for cancer initiating cells were identified, including CD34(+)/CD38(+) in leukemia, CD44(+)/CD24(+) in breast cancer, and CD133(+)/nestin(+) in brain tumor. Aberrant cell signal transduction pathway of stem cell is associated with malignant transformation, such as Wnt, Hedgehog, and Notch pathways. Up to our knowledge, the specific antigens expressed on ovarian cancer-initiating cells have not been identified and characterized yet. In the current study, using primary human ovarian tumors, the investigators will isolate and characterized ovarian cancer-initiating cells fully capable of reestablishing their original tumor hierarchy in vivo. The investigators will also elucidate the novel diagnostic and prognostic biomarkers on ovarian cancer-initiating cells by identifying numerous differentially potential surface antigens and/or over-expressed genes. Furthermore, a mouse ovarian cancer study model will be genetically engineered and investigated to monitor the possible therapeutic effects of immunotherapy and chemotherapy to these ovarian cancer-initiating cells. The investigators hope to specify and to stratify the molecular patterns, response to chemotherapy, prognostic biomarkers in patients with ovarian cancer-initiating cells. These results might offer some novel ovarian cancer therapy hypothesis to evaluate its function on tumorigenesis and potential on targeting ovarian cancer-initiating cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian carcinoma who undergo hysterectomy, bilateral oophorectomy and tubal resection, omentectomy, and appendectomy will be enrolled and the clinical data will be obtained from our hospital.

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | From disease diagnosis to death (Generally 2~5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan